CLINICAL TRIAL: NCT06586983
Title: Decentralization of Hepatitis B Care in Sub-Saharan Africa: a Pilot Program in Ethiopia
Status: Recruiting | Type: Observational
Sponsor: Oslo University Hospital (Other)
Collaborators: Norges ForskningsrÃ¥d, Stenberggata 26, pb. 2700, N-0131 Oslo, Norway (Unknown); Addis Ababa University (Other); Sykehuset i Vestfold HF (Other); St. Paul's Hospital Millennium Medical College, Ethiopia (Other)
Responsible Party: Principal Investigator, Asgeir Johannessen, Researcher / project manager, The Hospital of Vestfold
Other Study IDs: 656480
Record Dates: First submitted 2024-09-04; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Hepatitis B
Keywords: Liver cirrhosis; Antiviral agents; Liver disease; Resource-limited settings
MeSH Terms: conditions — Hepatitis B; Liver Cirrhosis; Liver Diseases | interventions — Tenofovir

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Dried blood spots
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Standard model ("treat only if"): HBsAg positive patients will be eligible for treatment of they fulfill one of the following criteria:
  i) Clinically diagnosed cirrhosis; or ii) APRI ≥0.5; or iii) Persistently elevated ALT >40 U/L; or iv) Co-infection with HCV or HDV; or v) Family history of HCC/cirrhosis; or vi) Relevant co-morbidity
  Interventions: Drug: Tenofovir Disoproxil Fumarate
- Inclusive model ("treat all except"): HBsAg positive patients will receive treatment, except if APRI ≤0.3 and no clinical signs/symptoms of cirrhosis and no risk factors for liver disease.
  Interventions: Drug: Tenofovir Disoproxil Fumarate
- Test-and-treat model ("treat all"): All HBsAg positive patients will receive treatment.
  Interventions: Drug: Tenofovir Disoproxil Fumarate

INTERVENTIONS:
Drug: Tenofovir Disoproxil Fumarate — 300 mg po OD

SUMMARY:
The goal of this observational study is to study models of care for decentralized hepatitis B treatment in Ethiopia.

Three different models of decentralized HBV care (standard model, simplified model, test-and-treat model) will be implemented at primary hospitals or health clinics in Ethiopia. Treatment will be given for free to patients who meet the treatment criteria. We will compare clinical outcome, laboratory outcomes and programmatic outcome measures between the 3 models.

DETAILED DESCRIPTION:
Chronic hepatitis B (CHB) is a major health problem globally, and in Ethiopia 5-10 % of the general population are infected with hepatitis B. In the absence of treatment, 15-40 % of these will die from its complications. Antiviral therapy effectively prevents disease progression and death in CHB. However, In low-income countries antiviral treatment is rarely available due to complex treatment guidelines, poor laboratory capacity, restrictions on antiviral treatment and lack of public funding.

In 2015, we set up a pilot treatment program for CHB at a tertiary hospital in Addis Ababa, Ethiopia. In 2021/22, this program was extended to four regional secondary hospitals to study simplified CHB care in a low-income country. With the present study we aim to decentralize CHB therapy to rural settings, which will be essential to achieve universal access to antiviral therapy in Africa. We will study different treatment models, each of which has its theoretical pros and cons: i) standard model ("treat only if…"), ii) inclusive model ("treat all except…"), and iii) test-and-treat ("treat all"). The primary endpoint will be death or liver decompensation, and secondary endpoints will be programmatic and laboratory success indicators. Moreover, we will study the cost-effectiveness of these decentralized models and compare with the tertiary/secondary hospital-based model.

Implementation research, such as our study, is of vital importance to respond to the research gaps identified by the World Health Organization in hepatitis B care. Our study is expected to directly inform international hepatitis B guidelines and will be a major contribution to the efforts to eliminate viral hepatitis as a public health threat by 2030.

ELIGIBILITY:
Inclusion Criteria:

* Adult (at least 18 years of age) who is HBsAg positive.

Exclusion Criteria:

* Below 18 years of age.
* Negative HBsAg rapid test at screening visit.
* Other disease with short life expectancy (disseminated cancer etc.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adults with a positive HBsAg rapid test are eligible for inclusion.
Sampling Method: Non-Probability Sample
Enrollment: 4500 (Estimated)
Dates: Start 2024-09-04 (Actual); Primary Completion 2028-09-05 (Estimated); Study Completion 2028-09-05 (Estimated)

PRIMARY OUTCOMES:
Death or liver decompensation | 3 years
  Deaths will be verified by tracing patients who miss appointments. Liver decompensation will be detected clinically and with liver function test assessed every 6-12 months.

SECONDARY OUTCOMES:
Linkage to care | 3 years
  Proportion of HBsAg positive patients on community screening that are linked to treatment center.
Loss to follow-up | 3 years
  Proportion of patients lost from care despite attempts of tracing patients who misses appointments.
Viral suppression | 3 years
  Proportion of patients with viral suppression, measured by HBV DNA test after 3 years in patients who receive treatment.
HIV incidence | 3 years
  Proportion of patients with deteced HIV infection during the 3 year follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Asgeir Johannessen, MD PhD, Study Director — The Hospital of Vestfold; Nega Berhe, MD PhD, Principal Investigator — Addis Ababa University
Locations (1):
- Addis Ababa University, Addis Ababa, Addis Ababa, Ethiopia

IPD SHARING:
Plan to Share IPD: Undecided
We don't intend to share IPD beyond our study group. However, the consent form describes sharing of IPD and we might consider this in the future if there are good scientific rationale to do so.